CLINICAL TRIAL: NCT06797947
Title: Describing the Clinical-laboratory Aspects of Diabetes by Creating a Registry in Which to Census All Newly Diagnosed or Already Diagnosed Cases After 1/1/2000 at the Endocrinology and Diabetes Prevention and Treatment Unit
Brief Title: Describing the Clinical-laboratory Aspects of Diabetes Through the Creation of a Registry
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: REDIA
Record Dates: First submitted 2024-12-03; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 29 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main objective of the study is to describe the clinical-laboratory aspects of diabetes by creating a registry in which to census all newly diagnosed or already diagnosed cases after 1/1/2000 at the O.U. of Endocrinology and Diabetes Prevention and Care.

DETAILED DESCRIPTION:
The main objective of the study is to describe the clinical-laboratory aspects of diabetes by creating a registry in which to census all newly diagnosed or already diagnosed cases after 1/1/2000 at the O.U. of Endocrinology and Diabetes Prevention and Care.

The clinical-laboratory aspects covered by this study also include family history, survival, comorbidities, psychological aspects, and in any case all those data that add relevant scientific information. This registry may be used to review the OU's case history and to confirm or obtain new scientific evidence on diabetes through cohort studies conducted using the data that will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Newly or previously diagnosed patients with diabetes mellitus at any stage of disease
* Obtaining informed consent

Exclusion Criteria:

- Patients whose diagnosis of diabetes mellitus is uncertain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation in the study will be offered consecutively to each patient with newly diagnosed diabetes mellitus evaluated at theU.O. of Endocrinology and Diabetes Prevention and Care.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2050-12-30 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical-Laboratory Aspects of Diabetes - Family History | through study completion, an average of 26 years
  This outcome measure will document and analyze the family history of diabetes in separate assessments:
  Diabetes in First-Degree Relatives: Data will be collected on the presence or absence of diabetes in parents, siblings, and offspring. This will be documented as a binary variable (yes/no) for each relative and reported as percentages of participants with affected first-degree relatives.
  Diabetes in Extended Family: Information will be collected on the presence of diabetes in second-degree and more distant relatives. This data will be categorized into groups based on the degree of relation and summarized descriptively as percentages of participants with a family history in extended relatives.
Clinical-Laboratory Aspects of Diabetes - Survival | through study completion, an average of 26 years
  This outcome measure will assess patient survival data, including:
  Overall Survival (OS): Defined as the time from study enrollment to death from any cause, reported in months.
  Life-Threatening Complications: Documented as binary outcomes (yes/no) and categorized by type (e.g., cardiovascular, respiratory).
  Each parameter will be recorded and analyzed separately:
  Survival status will be evaluated using Kaplan-Meier survival curves and summarized as median survival time with 95% confidence intervals.
  Complications will be reported as incidence rates (%) with descriptive statistics.
  Clinical and laboratory findings will be analyzed in separate measures to ensure clarity and avoid overlapping Units of Measure.
Clinical-Laboratory Aspects of Diabetes - Comorbidities | through study completion, an average of 26 years
  This outcome measure focuses on the presence of comorbid conditions among participants. The following comorbidities will be assessed:
  Hypertension: Documented as a binary variable (present/absent), based on clinical diagnosis and/or medication use.
  Cardiovascular Disease: Recorded as a binary variable (present/absent), categorized based on clinical diagnosis (e.g., coronary artery disease, heart failure).
  Kidney Disease: Assessed as a binary variable (present/absent), with relevant laboratory test results (e.g., eGFR in mL/min/1.73m²).
  Each comorbidity will be analyzed separately, reported as a percentage of participants with the condition, and presented with its respective unit of measurement (e.g., eGFR in mL/min/1.73m² for kidney disease). No aggregation of these conditions will occur within a single measure; each will be reported individually to ensure clarity.
Psychological Factors in Diabetes Management: Depression, Anxiety, and Quality of Life | through study completion, an average of 26 years
  This outcome measure will evaluate psychological factors related to diabetes management and well-being using specific, validated tools.
  Each of these psychological aspects will be assessed separately, with their corresponding scales and Units of Measure, to ensure clear reporting and analysis.
Blood Glucose and HbA1c Levels in Diabetes | through study completion, an average of 26 years
  This outcome measure will collect laboratory data on blood glucose and HbA1c levels:
  Blood Glucose Levels: Measured in mg/dL, collected as fasting blood glucose or postprandial glucose, reported as means ± standard deviation.
  HbA1c: Measured in percentage (%), summarized as mean ± standard deviation. These parameters will be analyzed independently to assess their role in diabetes management and outcomes.
Aggregated Data on Diabetes Progression and Management | through study completion, an average of 26 years
  This outcome measure will aggregate data collected from the diabetes registry, focusing on the following specific parameters:
  Diabetes-related Clinical Outcomes: These include metrics such as HbA1c levels (measured in %) and fasting blood glucose (measured in mg/dL), recorded at baseline and during follow-up visits.
  Comorbidities: Data on the presence of diabetes-related comorbidities, including hypertension (measured as systolic/diastolic blood pressure in mmHg) and cardiovascular events (binary variable: present/absent).
  Medication Use: Types and dosages of diabetes-related medications (e.g., insulin units, oral hypoglycemic agents), reported as frequencies or percentages.
  The aggregated data will be used to analyze trends in diabetes progression and management, summarized with descriptive statistics (mean ± standard deviation, percentages). The dataset will also be used for cohort studies to generate new scientific insights or validate existing evidence on diabetes.
Lipid Profile in Diabetes | through study completion, an average of 26 years
  This outcome measure will collect data on the lipid profile in patients with diabetes:
  Cholesterol (Total, HDL, LDL): Measured in mg/dL. Triglycerides: Measured in mg/dL. Data will be summarized as means ± standard deviation for each lipid component, with analysis focused on how these markers influence diabetes outcomes.
Kidney Function Tests in Diabetes | through study completion, an average of 26 years
  This outcome measure will collect laboratory data on kidney function in diabetes patients:
  Creatinine Levels: Measured in mg/dL. Estimated Glomerular Filtration Rate (eGFR): Calculated based on creatinine levels, age, gender, and race, expressed in mL/min/1.73m².
  Urinary Albumin-to-Creatinine Ratio (ACR): Measured in mg/g. These kidney function parameters will be reported independently to assess renal health in diabetes management.

CONTACTS AND LOCATIONS:
Overall Officials: Uberto Pagotto, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy